CLINICAL TRIAL: NCT03605823
Title: Pars Plana Ex-Press Mini Shunt for Management of Persistent Glaucoma in Vitrectomized Eye. A Potential Novel Technique.
Brief Title: Pars Plana Ex-Press Shunt in Vitrectomized Eyes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, abdussalam abdullatif, MD, Principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0123
Record Dates: First submitted 2018-07-23; First posted 2018-07-30 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma Secondary
Keywords: Express Mini shunt; Pars plana; Vitrectomized eye

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Express Mini shunt — Implantation of Express Mini shunt through pars plana in vitrectomized eyes

SUMMARY:
Implantation of Ex-Press Minishunt via the pars plana in treatment of secondary glaucoma in vitrectomized eyes achieves promising results avoiding complications of other surgical modalities.

DETAILED DESCRIPTION:
Ex-Press valve implantation was performed under peribulbar anesthesia (5 mL solution of 2% lidocaine and 2.5 mL of 0.5% bupivicaine [Marcaine]). A fornix-based conjunctival flap was dissected with a conjunctival incision made 2mm from the superior limbus and blunt dissection in the sub-Tenon space. Corneal tractional suture using 7-0 Vicryl was taken for proper exposure then gentle cautery was performed. A 4 × 3 mm × 2/3 the scleral thickness scleral flap was dissected at 11 o'clock centered on a point 3.5mm from limbus.

A cellulose microsponge soaked in 0.4 mg/mL Mitomycin-C solution was applied to the scleral flap, with the conjunctiva draped over the sponge for 3 minutes. The sponge was then removed and the area was washed with irrigating saline solution.

Using a pressure plate for globe fixation and as a measure, three 23G valved vitrectomy cannulae were inserted in the superonasal, superotemporal and inferotemporal quadrants. The superior peripheral retina was examined by indentation to ensure absence of any vitreous and more shaving is done at this area if residual vitreous was seen.

The scleral flap was lifted. With the infusion on, a 25-gauge needle was inserted in the scleral bed 3.5 mm from the limbus, through the pars plana into the vitreous cavity. The direction of insertion should be perpendicular to the scleral bed towards the mid-vitreous cavity. The needle was then removed. There must not be any lateral movement of the needle as this will cause aqueous to flow around the implant. The Ex-Press ® P50 shunt is preloaded on an injector and metal rod is fitted into the lumen of the shunt, attached to the end of the injector. The shunt was then placed through the ostium created with the needle. The angle of entry with the shunt was the same as the angle used to make the ostium. The shunt was rotated 90° so that it enters the eye with the spur facing the long axis of the entry point then it was inserted all the way into the wound followed by rotation to its final position once it is inside the eye so that the external backplate was flush with the scleral bed. The injector has an area on the shaft that was then depressed which retracts the metal rod in the lumen of the shunt. This allows the injector to be free from the lumen of the shunt.

After ensuring proper position of the shunt by examining it from inside the vitreous cavity with indentation, the two superior cannulae were removed and 7-0 Vicryl sutures were taken to ensure the water tightness of the sclerotomies.

The scleral flap was then sutured in place using two 10-0 nylon sutures with a spatulated needle. The tightness of the second suture was adjusted so that there was a good percolation with infusion pressure maintained at 15 mmHg in the vitrectomy machine settings. The last cannula together with the infusion was removed and the sclerotomy was sutured. IOP was adjusted to be between 10 mmHg and 20 mmHg. The conjunctiva was then meticulously closed with running 7-0 Vicryl suture in a watertight fashion. A fluorescein strip was used to make sure the wound was watertight.

During the six postoperative weeks, topical corticosteroids and antibiotics were administered four times a day.

ELIGIBILITY:
Inclusion Criteria:

* Secondary Glaucoma after vitrectomy not responding to maximum medical treatment

Exclusion Criteria:

* Phakic eyes
* Siliconized eyes
* History of Uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure control (IOP) | 6 month
  IOP less than 18 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No